CLINICAL TRIAL: NCT01931449
Title: Evaluation of a Modified Procedure of Digestive Tract Reconstruction Following Pancreatoduodenectomy: A Multicenter Randomized Controlled Study
Brief Title: Evaluation of A New Digestive Reconstruction Procedure Following Pancreatoduodenectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Huai-zhi Wang, Doctor, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NDR-2014-01
Record Dates: First submitted 2013-08-21; First posted 2013-08-29 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Pancreatic Cancer; Periampullary Carcinoma
Keywords: Pancreatoduodenectomy; Digestive Tract Reconstruction; Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modified digestive reconstruction (Experimental): Modified method of digestive tract reconstruction: Evaluate the resectability; Remove pancreas head, gastric pyloric antrum, duodenum, distal common bile duct and regional lymph nodes; Reconstruct digestive tract with an independent intestinal loop and pancreas end.
  Interventions: Procedure: Modified method of digestive tract reconstruction
- Routine pancreatoduodenectomy (Active Comparator): Routine digestive tract reconstruction: Evaluate the resectability; Remove pancreas head, gastric pyloric antrum, duodenum, distal common bile duct and regional lymph nodes;Reconstruct the common bile duct-jejunum and pancreatic duct-jejunum respectively.
  Interventions: Procedure: Routine digestive tract reconstruction

INTERVENTIONS:
Procedure: Modified method of digestive tract reconstruction
  Arms: Modified digestive reconstruction
Procedure: Routine digestive tract reconstruction
  Arms: Routine pancreatoduodenectomy

SUMMARY:
The purpose of this study is to evaluate the validity and safety of a modified operative procedure of digestive tract reconstruction following pancreatoduodenectomy which enables the pancreatic juice and bile to bypass at the pancreatointestinal anastomosis and merge at gastrointestinal anastomosis. It is anticipated that this procedure can decrease the risk of post-surgical pancreatic leakage and preserve the patients' digestive function as well.

DETAILED DESCRIPTION:
Pancreatoduodenectomy (PD) is one of the most complicated surgeries in abdominal clinical practice. It is widely used in the treatment of pancreatic head carcinoma, periampullary carcinoma, chronic pancreatitis with intractable pain, pancreatic head mass which unable to rule out pancreatic cancer. PD was improved in many ways in the last 80 years and the post-surgical mortality has decreased under 5%. Since the resected region of PD is wide including gall bladder, billiary tract, duodenum, pancreas, stomach, jejunum and regional lymph nodes. It has a high prevalence of complications, of which pancreatic leakage is the most common and serious one with a prevalence rate of 5-25% and mortality rate 20-50%。 The objective of the present study is to evaluate a new surgical procedure used for the digestive tract reconstruction following PD. The new procedure enables the pancreatic juice and bile to bypass at the pancreatointestinal anastomosis and merge at gastrointestinal anastomosis which can decrease the risk of post-surgical pancreatic leakage and keep the digestive function of patients. A multicenter, randomized, controlled study is designed to observe the prevalence of pancreatic leakage, other post-surgical complications, hospital stay, medical costs, life quality and other indexes to evaluate the efficacy and safety of this procedure. It is anticipated that through the study, this new procedure can be systematically verified if it is an ideal procedure of digestive reconstruction following PD which can be promoted into wider use.

ELIGIBILITY:
Inclusion Criteria:

* Below 80 years old
* CT (Computed Tomography), CTA (Computed Tomographic Angiography), MRI (Magnetic Resonance Imaging) or ultrasonic test suggested pancreatic head carcinoma, periampullary carcinoma, chronic pancreatitis with intractable pain, pancreatic head mass which unable to rule out pancreatic cancer, with or without obstructive jaundice/chronic abdominal pain.

Exclusion Criteria:

* Liver Metastasis
* Metastasis in common bile duct and hepatic duct
* Extensive lymph node metastasis, metastasis at hepatic portal or above pancreas
* Pancreatic head or periampullary has tight adhesion with postcava or aorta
* Distant metastasis
* Poor physical condition to tolerate anesthesia and surgery (e.g. severe cardio-pulmonary diseases, blood coagulation disorders)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Pancreatic Leakage | up to 12 months

SECONDARY OUTCOMES:
Life Quality Score | up to 12 months
Amylase Test of Abdominal Drainage Fluid | up to 3 months

OTHER OUTCOMES:
Anesthesia Score | up to 12 months
Length of Hospital Stay | up to 12 months
Re-surgery Rate | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Huai-zhi Wang, M.D., Ph.D., Principal Investigator — Southwest Hospital, China
Locations (1):
- Institution of Hepatobiliary Surgery, Southwest Hospital, Chongqing, Chongqing Municipality, China